CLINICAL TRIAL: NCT01112553
Title: Evaluation of Brain Activation in Complete Responders and Partial Responders Following Acute Administration of Treximet (Sumatriptan and Naproxen)
Brief Title: Treximet Migraine Brain Imaging Research Study
Acronym: TREX
Status: Terminated | Type: Observational
Why Stopped: Study was closed due to low enrollment numbers.
Sponsor: Mclean Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, David Borsook, MD, PhD, Senior Research Associate, Mclean Hospital
Other Study IDs: 2009-P-002689; 400483 (Other Grant/Funding Number: GlaxoSmithKline)
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Acute Migraine
Keywords: Acute Migraine; Treximet; Imaging; fMRI; Pain; Heat Stimulus
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Seven 5-mL blood samples will be drawn throughout the MRI session, and blood plasma will be analyzed for the concentration of Treximet.

GROUPS / COHORTS (1):
- Treximet: All migraine subjects will receive Treximet during a migraine episode at Visit 2.

SUMMARY:
We are looking for volunteers who suffer from acute migraine (<14 episodes per month) to participate in a 2-visit brain imaging research study. The goal of the study is to observe the effect of acute administration of Treximet during a migraine episode on the pain pathways of the migraine brain. Visit 1 will consist of 1 hour, where participants will be signing the informed consent form, completing questionnaires, meeting with the study physician, and having QST (sensory testing to determine individual pain thresholds to a heat stimulus) performed. Visit 2 will occur during a migraine episode. Volunteers will be asked to contact the study team at the first onset of a migraine. Upon arrival at Visit 2, individuals will be given an IV for blood draws. Once these the IV is in place, subjects will enter the MRI and be asked to stay very still. Scanning will occur for about 20 minutes, and then subjects will be given a Treximet tablet to combat their migraine. More scanning will follow Treximet administration. Some scans will have no stimulation, and others will apply a heat stimulus that subjects will rate using a pain scale. Seven 5-mL blood samples will be drawn throughout the duration of the MRI session. Both Visit 1 and Visit 2 will be compensated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (not pregnant or nursing)
* Age 18-65; with a focus on age 30-40 years
* Episodic migraine (experience migraine headache <14 days out of the month), with focus on left-sided pain
* Currently taking Treximet routinely for migraine treatment
* No significant medical history (No illnesses such as seizure disorder, diabetes, alcoholism, cardiac disease including coronary artery disease, psychiatric problems; drug addiction, respiratory problems, liver disease, etc.)
* No significant medication history, except for migraine
* Weight, <285 pounds
* Not claustrophobic
* No contraindication to taking triptans

Exclusion Criteria:

* Age <18 or > 65
* Significant medical problems (aside from pain before, during and after migraine episodes)
* Positive drug of abuse screen (excluding medications currently prescribed for their clinical condition, e.g. opioids, benzodiazepines, etc.)
* Use of opioid medications
* Claustrophobia
* History of dermatological hypersensitivity in the facial area
* Pregnancy
* Sensory loss detected on Quantitative Sensory Testing at screening
* Significant alcohol history (ingestion of 5 or more glasses (> 40 oz) of alcohol per week)
* Metal implants of any type (including dental bridges, crowns, retainers, orthodontic devices e.g. braces, etc.)
* Tattoos containing metallic ink on the neck, shoulders, upper arm and head (which could become heated up in the scanner, and potentially cause blistering or burning)
* Cardiac pacemakers
* Aneurysm clips and other vascular stents, filters, clips or other devices
* Prosthetic heart valves
* Other prostheses
* Neuro-stimulator devices
* Implanted infusion pumps
* Cochlear (ear) implants
* Ocular (eye) implants or known metal fragments in eyes
* Exposure to shrapnel or metal filings (sheet metal workers, welders, and others)
* Other metallic surgical hardware in vital areas
* Any known allergic side effects to Treximet
* Use of any of the following medications:
* Monoamine Oxidase A- Inhibitors (Azilect, Eldepryl, Marplan, Nardil, Parnate, Zelapar)
* SSRI's: citalopram/ Celexa, Lepraxo, paroxetine/ Paxil, fluoxetine/ Prozac, Sarafem, Symbyax, Sertraline/ Zoloft, Fluvoxamine/ Luvox
* SNRI's: duloxetine/ Cymbalta, venlafaxine/ Effexor
* Triptans: sumatriptan/ Imitrex, naratriptan/ Amerge, zolmitriptan/ Zomig, rizatriptan/ Maxalt, eletriptan/ Relpax, almotriptan/ Axert
* Ergotamine type medicines: Bellergal, Cafergot, Ergomar, Wiraine, Migranal/ DHE45, Sansert

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: English-speaking males or females between the ages of 18 and 65, who suffer from acute migraine (<14 migraine episodes/ month), will be recruited for this study.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2010-04; Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Borsook, MD, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- Neuroimaging Center, McLean Hospital, Belmont, Massachusetts, United States